CLINICAL TRIAL: NCT06809153
Title: Promoting Parallel Parenting: Putting Children First During High-Conflict Divorce and Separation (PCF)
Brief Title: Putting Children First - Parent Training for Parents in High Conflict
Acronym: PCF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRIS Media Inc (Other)
Responsible Party: Principal Investigator, Jordan Pennefather, Senior Scientist, IRIS Media Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R44HD111084-01A1 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Parenting Behavior; Parent Management Training; Parent-Child Relations; Child Behavior
Keywords: Online App
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: Two-arm design comparing the new intervention (PCF) to a business-as-usual control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Putting Children First (Experimental): Participants will be given access to the PCF app for 15 weeks.
  Interventions: Behavioral: Putting Children First
- Control - Business as Usual (No Intervention): Business as usual control participants will not be directed to any additional parenting trainings.

INTERVENTIONS:
Behavioral: Putting Children First — An online parenting intervention for families experiencing high inter-parental conflict during divorce or separation. Children in these families are at greater risk of adverse health outcomes such as mental illness, substance use, and social adjustment problems. Putting Children First will include evidence-based parent training and employ motivational interviewing to increase engagement, will promote parallel parenting to help parents minimize conflict, thereby mitigating negative health outcomes in their children.
  Arms: Putting Children First

SUMMARY:
Intervention efficacy will be evaluated via a randomized controlled trial in Indiana over 17 weeks with 250 dyads (i.e., divorcing/divorced/separated parents). Dyads will be randomized to business as usual (BAU) or BAU+PCF.

Compared to BAU, BAU+PCF will (a) increase parental self-efficacy, (b) decrease parental stress, (c) increase parental knowledge, (d) increase parental motivation to engage with the intervention, (f) increase the quality of parent-child relationships, and (g) improve parent-reported child stress and prosocial behaviors.

Parents with higher levels of conflict will be more responsive to parallel parenting, and increased parallel parenting among HIC dyads will lead to reductions in child adjustment problems.

DETAILED DESCRIPTION:
Intervention efficacy will be evaluated via a randomized controlled trial in Indiana over 17 weeks with 250 dyads (i.e., divorcing/divorced/separated parents). Dyads will be randomized to business as usual (BAU) or BAU+PCF. Given Indiana rules requiring parent education among divorcing and separating parents (i.e., BAU), the investigators expect nearly all divorcing parents to complete some form of parent education. Thus, the investigators will collect information from the court system on courses provided, as well as ask participants about the courses they have engaged in and the time spent. This aligns with best practice standards defining the control condition135; 136 and allows for a demonstration of whether PCF has benefits above and beyond existing interventions (BAU). The time spent on trainings will be included in the outcome analyses as a covariate. The trial will include 1 week for pre-test assessments, 9 weeks for PCF training, 6 weeks for reflection/practice, and 1 week for post-test assessments).

Hypotheses. The investigators hypothesize that:

Compared to BAU, BAU+PCF will (a) increase parental self-efficacy, (b) decrease parental stress, (c) increase parental knowledge, (d) increase parental motivation to engage with the intervention, (f) increase the quality of parent-child relationships, and (g) improve parent-reported child stress and prosocial behaviors.

Parents with higher levels of conflict will be more responsive to parallel parenting, and increased parallel parenting among HIC dyads will lead to reductions in child adjustment problems.

Participants. The sample will consist of parents who have recently experienced (within the past 2 years) divorce or separation, or are currently divorcing or separating, and who have children aged 4-12. Parents will be referred to the PCF intervention from family courts in Indiana (see Letters of Support) as they are identified by the court system as experiencing HIC. To approximate the real world and ensure that the sample is representative, family court judges, who would likely mandate completion of this intervention, will refer families they deem "high conflict." To be eligible for the study, both parents must consent. Because the stress of divorce and high levels of conflict can be deleterious to mental health and well-being, all participants in the study will be provided with a list of resources for individuals experiencing mental health, substance use, or intimate partner violence in their local area, and will be encouraged to seek assistance if needed. Attrition rates of parenting interventions are often high.137 However, the investigators have instituted practices to enhance retention (e.g., regular reminders, reasonable pacing of the training to 1 module per week, motivational interviewing). From the investigators experience in similar studies, the investigators expect attrition of less than 30%.42; 138 Since the research design requires both members of the dyad to complete the assessments, the investigators define attrition as one parent failing to complete posttest assessments. The investigators plan to recruit 250 dyads (500 parents) to ensure a final sample of at least 175 dyads (see Power Considerations).

ELIGIBILITY:
Inclusion Criteria:

* parents who have recently experienced (within the past 2 years) divorce or separation, or are currently divorcing or separating.
* have children aged 4-12.
* Dyadic recruitment (both parents).
* identified by the court system as experiencing HIC.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Parenting Practices | Baseline and 15 weeks
  Parenting practices will be assessed using the Parenting Practices Inventory, a 72-item survey using a 4-point Likert-type scale with rating from 1 to 4 and higher scores indicating more use of the practice, thus higher scores are better outcomes. The subscales have demonstrated adequate internal reliability (alphas = .54 to .80) and have been used in multiple studies to evaluate parenting interventions
Parenting efficacy | Baseline and 15 weeks
  Parenting efficacy will be assessed using four, 6-item subscales from the Tool for Measuring Parent Self-Efficacy, measuring domains of play and enjoyment, discipline practices, perceived control in parenting, and acceptance of parenting role (internal consistency alphas = .80 to .89). Scores range from 1 "agree a lot" to 3 "don't know", with scores on the subscales ranging from 6 to 18 and higher scores indicating less self-efficacy, a worse outcome.
Parenting stress | Baseline and 15 weeks
  Parenting stress will be assessed using the Parenting Stress Scale, which is a brief 18-item Likert-type scale that includes four domains: parental rewards, parental stressors, lack of control, and parental satisfaction. Each item is on a 5-point scale ranging from 1 "Strongly Disagree" to 5 "Strongly Agree". The total scale (after reverse coding half the items) results in possible scores ranging from 18 to 90 with higher scores indicating more parenting stress. The scale has demonstrated good internal reliability (alphas = .86 to .88). This instrument is commonly used for both clinical and non-clinical samples.
Interparental conflict | Baseline and 15 weeks
  The Divorce Conflict Scale is a 6-item screener specifically addressing conflict and cooperation post-relationship/marital dissolution with good internal reliability (alpha reliability = .88). One item uses a 6 point scale ranging from 1 "all of the time" to 6 "at no time"; one item uses a 5-point scale ranging from 1 "very low level of conflict" to 5 "very high level of conflict"; the other 4 items use a 4-point Likert scale ranging from 1 "Strongly Agree" to 4 "Strongly Disagree". The total score ranges from 6 to 27, with higher scores indicating more conflict (worse outcome).
Motivation to engage with the PCF | Baseline and 15 weeks
  Motivation to engage with the Putting Children First training materials will be assessed using the Situational Motivation Scale. This is a 16-item Likert-type scale with four internally consistent factors (internal consistency alphas > .77): intrinsic motivation, identified regulation, external regulation, and motivation. It uses a 7-point Likert Scale ranging from 1 "does not correspond at all" to 7 "corresponds exactly". The averages for each subscale are calculated with higher scores indicating higher motivation (positive outcome). This measure has been used extensively to evaluate motivation in many contexts and towards many activities, including mandated training.
Child behavior - Strengths and Difficulties Questionnaire | Baseline and 15 weeks
  Parent reports of child behavior will be assessed using the Strengths and Difficulties Questionnaire a brief behavior rating scale for 3- to 16-year-olds that assesses functioning in five domains, each with five items: emotional symptoms (alpha = .80), conduct problems (alpha = .77), hyperactivity (inattention, alpha = .90), peer problems (alpha = .63), and prosocial behavior (alpha =.83).Internal consistency alpha estimates were based on Low et al. The Strengths and Difficulties Questionnaire uses a 3-point scale ranging from 0 "Not True" to 2 "Certainly True". Totals for each subscale are calculated, with higher scores on prosocial behaviors indicating a positive outcome and higher scores on the other four indicating negative outcomes.
Child Behavior - Eyberg Child Behavior Inventory | Baseline and 15 weeks
  The Eyberg Child Behavior Inventory is a 36-item scale completed by parents about their children's behavior (ages 2-16 years) at home using a 7-point Intensity scale and a yes-or-no Problem scale. It identifies conduct problems such as noncompliance, defiance, aggressiveness, and impulsiveness. The Intensity and Problem scales demonstrate good psychometrics, with high internal consistency (both scales alpha = .98), significant test-retest reliability. The subscale averages range from 1 to 7, with higher scores indicating higher levels of negative child behavior.

IPD SHARING:
Plan to Share IPD: Yes
We will provide de-identified data for additional analysis to any qualified individual in the scientific community.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the final report of the grant is submitted and associated publications are accepted we will make the de-identified final research data and associated codebooks available within 6 months.